CLINICAL TRIAL: NCT05553327
Title: Impact of a Multimodal Prehabilitation Program Before Robotic-assisted Radical Prostatectomy. A Randomized Clinical Trial.
Brief Title: Impact of a Multimodal Prehabilitation Program Before Robotic-assisted Radical Prostatectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2021/0289
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group of patients will not receive a pre-hab program
- Multimodal prehabilitation (Experimental): This patients will receive the pre-hab program
  Interventions: Behavioral: Multimodal prehabilitation

INTERVENTIONS:
Behavioral: Multimodal prehabilitation — * Physical state: individualised physical status will be evaluated by a physiotherapist. A specific training program and pelvic floor exercises sessions will be led by a physiotherapist.
  * Nutritional state: individual nutritional status will be evaluated by a nutritionist and intervention will be done if applicable. A nutrition group session will be held.
  * Mental health: mindfulness group sessions led by psychologists will be held.
  Arms: Multimodal prehabilitation

SUMMARY:
The aim of the study is to verify whether a multimodal prehabilitation programme prior to robotic radical prostatectomy contributes to a faster recovery of quality of life after surgery, to better functional results (including erectile function and continence) and to less perioperative anxiety.

DETAILED DESCRIPTION:
Single center randomized clinical trial including prostate cancer patients undergoing robotic-assisted radical prostatectomy at the Hospital Clínic de Barcelona. Patients will be randomized into two groups, one receiving multimodal prehabilitation and the other a control group. Multimodal prehabilitation consists of improving the functional and mental capacity of an individual to cope with a significant stressor, in this case surgery. The design of our prehabilitation program, lasting 4 weeks prior to surgery, consists of three parts; physical state, nutritional state and mental health. In the case of physical condition, a series of supervised and "home-based" exercises (aerobic and functional) will be carried out in addition to specific pelvic floor exercises. The nutritional status will be evaluated by a nutritionist. Diet guidelines will be given and if there are deficiencies they will be supplemented. Regarding mental health, a visit will be made with a psychologist and group and online therapies will be offered. The outcomes will be evaluated before starting the prehabilitation program, at the end of it (just before surgery) and at 4, 8 and 16 weeks after surgery. The outcomes include variables on physical, nutritional and mental state, health-related quality of life (HRQoL), and continence and erectile function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized prostate cancer
* Candidates to robotic radical prostatectomy

Exclusion Criteria:

* Non-localized prostate cancer
* Previous history of pelvic radiotherapy or pelvic surgery
* Failure to consent,
* Unwillingness to participate
* Anticipated failure to adhere to the program sessions.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 100 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Continence recovery | Week 0 and 4 (pre-op); weeks 8, 16 and 28 (post-op)
  Change in continence during the prehabilitation program and postoperative recovery.
  International Consultation on Incontinence Questionnaire (ICIQ)
  Scoring scale: 0-21 Higher value means worse outcome
Perioperative anxiety levels | Week 0 and 4 (pre-op); weeks 8, 16 and 28 (post-op)
  Change in perioperative anxiety levels
  Hospital Anxiety & Depression (HAD )
  Scoring scale: 0-21 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)

SECONDARY OUTCOMES:
Change in physical status by STS | Week 0 and 4 (pre-op); weeks 8, 16 and 28 (post-op)
  Sit-to-Stand (STS)
  Time needed for 5 repeated chair rises. Higher time means worse physical status.
Change in physical status by 6MWT | Week 0 and 4 (pre-op); weeks 8, 16 and 28 (post-op)
  6 Minute Walk Test (6MWT)
  Distance covered over a time of 6 minutes. Higher time means worse physical status.
Change in perception of physical status | Week 0 and 4 (pre-op); weeks 8, 16 and 28 (post-op)
  Yale physical activity survey (YPAS)
  Part 1 - Scoring scale: 0-85680 kcal/week Part 2 - Scoring scale: 0-142 Part 3 - Scoring scale: 0.7-1.3
  Higher values indicates higher activity.
Erectile function recovery | Week 0 and 4 (pre-op); weeks 8, 16 and 28 (post-op)
  International Index Erectile Function (IIEF-5)
  Change in erectile function during the prehabilitation program and postoperative recovery.
  Scoring scale: 5-25 22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction
Change in perceived general quality of life | Week 0 and 4 (pre-op); weeks 8, 16 and 28 (post-op)
  EORTC QLQ - C30
  Scoring scale: 0-100 Higher value indicates higher perceived general quality of life
Change in perceived prostate quality of life | Week 0 and 4 (pre-op); weeks 8, 16 and 28 (post-op)
  EORTC QLQ - PR25
  Scoring scale: 0-100 Higher value indicates higher perceived prostate quality of life
Early postoperative morbidity by CDC | Week 8 (post-op)
  Clavien-Dindo Classification (CDC)
  Scoring scale: 1-5 Higher value indicates more severe complication
Early postoperative morbidity by CCI | Week 8 (post-op)
  Comprehensive Complications Index (CII)
  Scoring scale: 0-100 Higher value indicates more severe complication
Perceived application usability | Week 4
  Usability questionare
  Includes a combination of the System Usability Scale (SUS) and the Net Promoter Score (NPS).
  Scoring scale: 0-100 Higher value indicates better perceived usability
Satisfaction with the multimodal program | Week 4
  Satisfaction questionnaire
  Scoring scale: 0-45 Higher value indicates higher satisfaction
Nutritional status | Week 0 and 4
  Nutritionist final evaluation summarized as optimal or suboptimal by the specialist.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Vilaseca, Dr, Principal Investigator — Clinic
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No